CLINICAL TRIAL: NCT04675060
Title: A Study of the Effect of High-fat Meal on the Pharmacokinetics of Oral TQ-B3139 Capsules in Patients With Solid Tumor
Brief Title: Effect of High-fat Meal on the Pharmacokinetics of TQ-B3139 Capsules
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3139-I-02
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): TQ-B3139 capsules administered single dose of 600 mg under fasted conditions in day 1 followed by single dose of 600 mg with a high-fat meal in day 5, then TQ-B3139 capsules administered 600mg orally, twice daily.
  Interventions: Drug: TQ-B3139 capsules
- Cohort 2 (Experimental): TQ-B3139 capsules administered single dose of 600 mg with a high-fat meal in day 1 followed by single dose of 600 mg under fasted conditions in day 5, then TQ-B3139 capsules administered 600mg orally, twice daily.
  Interventions: Drug: TQ-B3139 capsules

INTERVENTIONS:
Drug: TQ-B3139 capsules — TQ-B3139 capsules administered 600mg orally, twice daily in 28-day cycle.

SUMMARY:
This is a study to evaluate the effect of high-fat meal on the pharmacokinetics of TQ-B3139 capsules in patients with solid tumor

ELIGIBILITY:
Inclusion Criteria:

* 1. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 1.

  2. Life expectancy ≥12 weeks. 3. Patients with confirmed gene mutations, including ALK fusion, ROS1 fusion, MET mutation or amplification.

  4. Adequate organ system function. 5.Female patients of childbearing age should agree to use contraceptive measures during the study period and for at least 6 months after study is stopped; male patients should agree to use contraception during the study period and for at least 6 months after study is stopped.

  6.Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has other malignancies within 3 years. 2. Has multiple factors affecting oral medication. 3. The toxicity of previous antitumor treatment is not recovered to ≤ grade 1(CTCAE 5.0) .

  4. Has received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before the first dose.

  5. Has long-term unhealed wounds or fractures. 6. Has a history of psychotropic drug abuse or have a mental disorder. 7. Has any severe and/or uncontrolled disease. 8. Has received surgery, chemotherapy, radiotherapy or other anticancer therapies 4 weeks or 5 half-life of drug elimination (whichever comes first) before the first dose.

  9. Has participated in other clinical studies within 4 weeks before enrollment. 10.Using inhibitors or inducers of CYP3A at present. 11. Has receiving Chinese patent medicines with anti-tumor indications in the drug instructions that NMPA approved within 2 weeks before the start of the study treatment.

  12. Pleural effusion, pericardial effusion or ascites that cannot be controlled and need repeated drainage.

  13. Brain metastases with symptoms or symptoms of brain metastases were controlled for less than 2 weeks.

  14. In lactation period or plan to breastfeed during the study period. 15.According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | 0hour, 1hour, 2hour, 3hour, 4hour, 5hour, 6hour, 7hour, 8hour, 10hour, 24hour, 48hour,72hour, 96hour on day 1 and day 5.
  To characterize the pharmacokinetics of TQ-B3139 by assessment of area under the plasma concentration time curve from zero to time.
AUC0-∞ | 0hour, 1hour, 2hour, 3hour, 4hour, 5hour, 6hour, 7hour, 8hour, 10hour, 24hour, 48hour,72hour, 96hour on day 1 and day 5.
  To characterize the pharmacokinetics of TQ-B3139 by assessment of area under the plasma concentration time curve from zero to infinity.
Cmax | 0hour, 1hour, 2hour, 3hour, 4hour, 5hour, 6hour, 7hour, 8hour, 10hour, 24hour, 48hour,72hour, 96hour on day 1 and day 5.
  Cmax is the maximum plasma concentration of TQ-B3139 or metabolite(s).

SECONDARY OUTCOMES:
Tmax | 0hour, 1hour, 2hour, 3hour, 4hour, 5hour, 6hour, 7hour, 8hour, 10hour, 24hour, 48hour,72hour, 96hour on day 1 and day 5.
  To characterize the pharmacokinetics of TQ-B3139 by assessment of time to reach maximum plasma concentration.
t1/2 | 0hour, 1hour, 2hour, 3hour, 4hour, 5hour, 6hour, 7hour, 8hour, 10hour, 24hour, 48hour,72hour, 96hour on day 1 and day 5.
  t1/2 is time it takes for the blood concentration of TQ-B3139 or metabolite(s) to drop by half.
Objective Response Rate (ORR) | up to 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR).
Progression-free survival (PFS) | up to 24 months
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Disease control rate (DCR) | up to 24 months
  Percentage of participants achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Duration of response (DOR) | up to 24 months
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China